CLINICAL TRIAL: NCT03389217
Title: Efficacy of tDCS on Pain Experience in People With Multiple Sclerosis: A Pilot Randomized Control Trial
Brief Title: Efficacy of tDCS on Pain in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, Principal Investigator, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS_tDCS_Pain
Record Dates: First submitted 2017-11-16; First posted 2018-01-03 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Pain; Transcranial Direct Current Stimulation; tDCS
MeSH Terms: conditions — Multiple Sclerosis; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-tDCS + rehabilitation programme (Experimental): The real transcranial Direct Current Stimulation group will consist of anodal transcranial direct current stimulation applied for a total duration of 30 minutes over the the left dorsolateral prefrontal cortex and rehabilitation programme for prevention and management of pain.
  Interventions: Device: Real-tDCS + rehabilitation programme
- Sham-tDCS + rehabilitation programme (Active Comparator): The sham transcranial Direct Current Stimulation group will consist of anodal transcranial direct current stimulation applied for a total duration of 30 s over left dorsolateral prefrontal cortex and rehabilitation programme for prevention and management of pain.
  Interventions: Device: Sham-tDCS + rehabilitation programme

INTERVENTIONS:
Device: Real-tDCS + rehabilitation programme — tDCS stimulation will be delivered using a constant current stimulator, with rechargeable batteries. The active electrode will be placed on the left dorsolateral prefrontal cortex (DLPFC) and the reference electrode will be placed over the controlateral supraorbital region. The direct current will be delivered through a pair of sponge electrodes with a surface of 35 cm2 (7 × 5), soaked in saline solution. This continuous stimulation will last 30 minutes, with an intensity of 1 mA. Rehabilitation programme will last for 30 minutes and includes specific exercises for prevention and management of pain. All the subjects enrolled will receive treatments for 4 weeks. During the first week the experimental group underwent tDCS daily (Monday-Friday) and rehabilitation programme 3 days per week. tDCS will be delivered before rehabilitation treatment. During the second, third and fourth week subjects will receive only rehabilitation treatment, 3 days per week.
  Arms: Real-tDCS + rehabilitation programme
Device: Sham-tDCS + rehabilitation programme — The control group will receive the same protocol treatment but they underwent sham-tDCS during the first week of treatment. For sham condition tDCS, current was delivered for only 30 seconds and then the current was discontinued, but the tDCS apparatus was left in place for the same time as active tDCS (30 minutes)
  Arms: Sham-tDCS + rehabilitation programme

SUMMARY:
Pain is a common symptom experienced by people with MS and can significantly interfere with participation in the activities of daily living and adversely affect health-related quality of life. Pain in people with MS has the potential to become chronic, as a consequence of neuronal reorganization. Transcranial Direct Current Stimulation (tDCS) promotes the modulation of brain activity and its prolonged and continuous application can effect plastic modification. Combining tDCS with rehabilitation treatment may have effect in reducing pain in people with MS. This is a pilot randomized control trial to test the effects of tDCS in MS-related pain rehabilitation, its efficacy on pain (intensity, quality, interference with physical functioning), catastrophizing, emotional functioning and quality of life. Furthermore, we will explore the effects on pressure pain threshold and EEG recording. Correlations between sample characteristics and pain features will be investigated. Considering role of tDCS on neuropsychological functions, selective attention will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain defined as a constant or intermittent sensory symptom with unpleasant feelings or pain, lasting more than 3 months with a minimum score of 3 points on the Numeric Rating Scale (NRS) for pain perception;
* lack of MS worsening in the three months just before the intervention period;
* cognitive functioning to give informed consent identified by a Mini-Mental Status Examination (MMSE) score ≥ 24/30.

Exclusion Criteria:

* worsening of MS-related conditions or changes in drug therapy or any other confounding factor during the study;
* rehabilitation treatments or Botulinum toxin injections during the three months preceding the start of the study;
* intracranial metal implants that can be stimulated, incorrectly positioned, or overheated by the electric current;
* severe cardiopulmonary, renal, and hepatic diseases;
* pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | 4 weeks
  Core outcome measure of pain intensity in chronic pain treatments' clinical trials

SECONDARY OUTCOMES:
Short Form McGill Pain Questionnaire (SF-MPQ) | 1 week, 4 weeks, 8 weeks
  Assessment of sensory and affective dimensions of typical whole-body pain intensity.
Brief Pain Inventory (BPI) | 1 week, 4 weeks, 8 weeks
  Assessment of the extent to which pain interferes with general activity, mood, walking, work, relationship with others, sleep, and enjoyment of life.
Pain Catastrophizing Scale (PCS) | 1 week, 4 weeks, 8 weeks
  Assessment of a tendency to misinterpret or exaggerate apparently threatening situations that can lead to increased sensitivity to pain.
Coping Strategies Questionnaire (CSQ) | 1 week, 4 weeks, 8 weeks
  Assessment of the frequency of coping strategies in response to pain.
Beck Depression Inventory II (BDI-II) | 1 week, 4 weeks, 8 weeks
  Assessment of severity of common depressive symptoms.
MS Quality of Life - 54 (MSQOL-54) | 1 week, 4 weeks, 8 weeks
  Multidimensional health-related quality of life measure that combines both generic and MS-specific items
Fatigue Severity Scale (FSS) | 1 week, 4 weeks, 8 weeks
  Assessment of common features of fatigue in patients with multiple sclerosis
Go/No-go Task | 1 week, 4 weeks, 8 weeks
  Assessment of selective attention
Patient Global Impression of Change (PGIC) | 1 week, 4 weeks, 8 weeks
  Measure of participants' assessment of the clinical importance of their improvement or worsening over the course of a treatment
Pressure Pain Threshold (PPT) | 1 week, 4 weeks, 8 weeks
  PPT is measured to test presence of widespread pressure hyperalgesia as sign of abnormal pain processing.
Electroencephalography (EEG) recordings | 1 week, 4 weeks, 8 weeks
  EEG data will be recorded to test presence of particular brain activity in condition of pain chronicity and catastrophization.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Straudi, MD, PhD, Study Director — Ferrara Rehabilitation Hospital
Locations (1):
- Ferrara University Hospital, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No